CLINICAL TRIAL: NCT05191108
Title: The Effect of Mindfulness Stress Reduction Program on Premenstrual Symptoms: A Randomized Controlled Study
Brief Title: Premenstrual Syndrome (PMS) and Mindfulness Stress Reduction Program (MSRP)
Acronym: PMS and MSRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NURDİLAN SENER (Other)
Collaborators: Kırklareli University (Other)
Responsible Party: Sponsor-Investigator, NURDİLAN SENER, Assistant Professor, Firat University
Organization: Firat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Firat Universityyy
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Premenstrual Syndrome
Keywords: mindfulness; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomize Controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of mİNDFULNESS Stress Reduction Program on Premenstrual Symptoms (Experimental): In order to prevent bias in the study groups, the Introductory Information Form and PMSS scale will be applied via online Google forms. Participants who meet the criteria will be randomly assigned to the mindfulness stress reduction group (Group 1) and control group (Group 2) in the number determined by power analysis and a simple random number generator program (www.random.org). These experimental and control groups will be recorded by the researchers as a list. Participants participating in the study will be informed about the mindfulness stress reduction application, but they will not be informed about what the mindfulness stress reduction application does (single-blind method). These participants will be asked to sign the consent form by expressing that they can withdraw from the study at any time.
  Interventions: Behavioral: mindfulness stres reduction programe
- Control group (No Intervention): not routinely do anything to reduce premenstrual symptoms

INTERVENTIONS:
Behavioral: mindfulness stres reduction programe — Complaints about PMS and sharing information about these complaints, Practice of breathing focused meditation, mplementation of mindful eating exercises,Raising awareness in daily activities,Teaching the body scanning exercise and repeating this practice during the week with the audio recordings given.Ensuring environmental awareness Ensuring that you live by being aware of the moments experienced during the week, 20 minutes of sitting breathing focused sitting meditation Coping with stress Sharing the experiences of the previous week Implementation of mindful vision practices Explaining the relationship between stress and experienced events.Eating exercises Mindful breathing Ensuring environmental awareness Explaining the importance of thinking about the relationship between stress and their reactions and accepting them without judgment, and sharing the experiences at the end of the day of silence.
  Other Names: mindfulness
  Arms: The Effect of mİNDFULNESS Stress Reduction Program on Premenstrual Symptoms

SUMMARY:
Premenstrual syndrome (PMS) is a disorder characterized by emotional, physical and behavioral symptoms that increase the severity of the menstrual cycle in women of reproductive age during the luteal phase and disappear spontaneously a few days after the onset of menstruation. Nonpharmacological applications are often preferred to reduce premenstrual symptoms. It has been stated that with the meditation practices of mindfulness, individuals experience less anxiety, depression, anger and lower levels of psychological distress, including anxiety. . It is thought that the mindfulness stress reduction program can reduce the symptoms of PMS by regulating the stress level and emotional balance of women.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a disorder characterized by emotional, physical and behavioral symptoms that increase the severity of the menstrual cycle in women of reproductive age during the luteal phase and disappear spontaneously a few days after the onset of menstruation. It is stated in the literature that more than 40 million women experience PMS symptoms. While PMS significantly affects 20% of women's daily lives, it manifests itself as mild premenstrual symptoms in 90% of women. It is stated that PMS is associated with more than 300 physical, psychological, emotional, behavioral and social symptoms. These symptoms can include changes in appetite, weight gain, abdominal pain, backache, lower back pain, headache, breast swelling and tenderness, nausea, constipation, anxiety, irritability, anger, fatigue, restlessness, mood swings, and crying. Therefore, premenstrual symptoms can negatively affect individuals' participation in courses, school success, social activities and family relationships. Recently, in addition to pharmacological applications, non-pharmacological applications are frequently preferred to reduce premenstrual symptoms (reflexology, acupuncture, acupressure, music, mindfulness).

Mindfulness is defined as directing one's non-judgmental attention to thoughts, feelings, bodily sensations, and interactions. It has been stated that with the meditation practices of mindfulness, individuals experience less anxiety, depression, anger and lower levels of psychological distress, including anxiety. . PMS is an important health problem with complex symptoms. To cope with these symptoms, PMS needs to be addressed in a multidimensional way. It is thought that the mindfulness stress reduction program can reduce the symptoms of PMS by regulating the stress level and emotional balance of women. When the domestic studies were examined, there was no study that evaluated the effect of mindfulness stress reduction program on PMS, while when the foreign literature was examined, it was determined that there were studies conducted in a limited number and with a small sample, in which the effect of mindfulness stress reduction program on PMS was evaluated. This research was planned as a single-blind randomized controlled experimental study to evaluate the effect of mindfulness stress reduction program on the reduction of premenstrual symptoms in coping with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-30
* Having a score of 45 or more on the PMS scale
* Regular menstruation (between 21-35 days)
* Knowing Turkish (being literate)
* Read and approve the voluntary consent form

Exclusion Criteria:

* Having any gynecological disease (abnormal uterine bleeding, uterine fibroids, ovarian cysts, hormonal treatment, etc.),
* Having a chronic or physical illness (having serious hearing and vision problems, vestibular disorders that can cause balance loss)
* Having any problem that prevents communication (such as not knowing Turkish, having impairment in hearing, speaking and understanding abilities)
* Receiving a psychiatric treatment (Pharmacotherapy or psychotherapy)
* Do not use pharmacological or non-pharmacological applications to reduce the symptoms of premenstrual symptoms.

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — PMS IS ONLY SEEN IN WOMEN
Enrollment: 74 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
premenstrual syndrome | UP TO 16 WEEKS
  This scale, which was developed by Gençdoğan et al. (2006) for the evaluation of premenstrual symptom complaints, consists of 44 questions in total. The scale has nine sub-dimensions: depressive affect, anxiety, fatigue, irritability, depressive thoughts, pain, appetite changes, sleep changes, and swelling. PMSS is performed by evaluating the person retrospectively, taking into account the status of being "within 1 week before menstruation". The lowest score to be obtained from the scale is 44, and the highest score is 220. High scores indicate an increase in the intensity of PMS. In calculating the scale score, 44 points are considered as No PMS, 45-103 points as PMS Mild, 104-163 points as PMS Moderate, and 164-220 points as PMS Severe Level. Cronbach's α reliability coefficient is between 0.75 for the total scores of the scale and between 0.75 and 0.91 for the subscales. Written permission was obtained from Gençdoğan for the use of the scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - NURDİLAN, Elâzığ, Eyalet/Yerleşke
  - Kırklareli Üniversitesi, Kırklareli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sener Cetin N, Solt Kirca A. The Effect of a Mindfulness-Based Stress Reduction Program on Premenstrual Symptoms: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Sep-Oct;68(5):604-610. doi: 10.1111/jmwh.13530. Epub 2023 Jun 19. PMID 37335817